CLINICAL TRIAL: NCT06293859
Title: Effect of Daily Lactococcus Cremoris Spp. Consumption Immobilized in Oat Flakes on Blood and Urine Biomarkers and Human Microbiome: a Randomized Placebo-controlled Clinical Trial
Brief Title: Effect of 12-week Probiotic Consumption Immobilized on Oat Flakes on Blood and Urine Biomarkers and Human Microbiome
Acronym: FOODBIOMES CT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Aegean (Other)
Collaborators: Democritus University of Thrace (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5047292
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional oat flakes-placebo (Placebo Comparator)
  Interventions: Other: Conventional oat flakes
- Probiotic oat flakes (Experimental)
  Interventions: Other: Probiotic oat flakes

INTERVENTIONS:
Other: Probiotic oat flakes — 2 x 10^9 cfu/g Lactococcus cremoris immobilized on oat flakes
  Arms: Probiotic oat flakes
Other: Conventional oat flakes — Commercial oat flakes
  Arms: Conventional oat flakes-placebo

SUMMARY:
The purpose of this clinical trial was to evaluate the effects Lactococcus cremoris spp. im-mobilized on oat flakes on human microbiome and blood and urine biomarkers of associated with human health.

DETAILED DESCRIPTION:
All eligible and consenting individuals were assigned a unique code for identification purposes. They were then randomly assigned to either the probiotic or placebo group. The probiotic group received oat flakes containing immobilized Lactococcus cremoris, while the placebo group received oat flakes indistinguishable in color, smell, and taste from the flakes with immobilized probiotics.Participants received written instructions on storing the product, which required refrigeration. They were instructed to consume 5 g of oats daily with a meal, ensuring the meal's temperature remained below 35 °C and was non-acidic (e.g., with yogurt). Biological samples were collected at three time points; before intervention, at 6th and 12th week.

ELIGIBILITY:
Inclusion Criteria:

* participants to be aged between 18 and 65 years
* clinically tested with fasting plasma glucose less than 100 mg/dL
* clinically tested withcholesterol less than 220 mg/dL
* otherwise healthy

Exclusion Criteria:

* body mass index [BMI] higher than 40 kg/m2 (morbidly obese)
* following a diet plan for weight loss
* following a contraceptive treatment or taking probiotic supplements
* following medication with an effect on lipaemia or glycemia indicators
* having any allergies/intolerances to trial ingredients
* pregnant or planning to become pregnant or breast feeding
* users of illicit drug, having a chronic alcoholism or total daily alcohol intake more than 50 g per day
* diagnosed with a chronic condition (cancer, active liver disease, severe kidney dysfunction, severe stroke in the last six months and conditions associated with an increased risk of bleeding) or any other serious medical condition that may affect the individual's ability to participate in a dietary intervention study
* considered unreliable by the researcher or having a shorter life expectancy than the expected duration of the study due to some illness or if they were in any situation in which by the researcher's opinion their participation in the study was not considered safe (e.g. drug addiction, alcohol abuse).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers | Blood samples were collected by venipuncture at three time points; before intervention, at 6th and 12th week
  Change from baseline of hs-CRP and IL-6

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Aegean, Myrina, Limnos/Lesvos, Greece

IPD SHARING:
Plan to Share IPD: No